CLINICAL TRIAL: NCT01646554
Title: BOS3: Randomized Phase II/III Trial Evaluating the Efficacy of FOLFOX Alone Versus FOLFOX Plus Aflibercept in K-ras Mutant as Perioperative Treatment in Patients With Resectable Liver Metastases From Colorectal Cancer.
Brief Title: Efficacy of FOLFOX Versus FOLFOX Plus Aflibercept in K-ras Mutant Patients With Resectable Liver Metastases
Acronym: BOS3
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1207; 2012-002317-18 (EudraCT Number)
Record Dates: First submitted 2012-07-16; First posted 2012-07-20 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Cancer Metastatic; Liver Metastases; KRAS Mutated Colorectal Cancer
Keywords: Liver metastases; Colorectal Cancer; KRAS mutated; FOLFOX; Aflibercept; Randomized; Phase II-III; Perioperative treatment; Adjuvant; Neo-adjuvant; Surgery; Progression Free Survival
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; aflibercept; Surgical Procedures, Operative

ARMS (2):
- Arm A: modified FOLFOX6 and Surgery (Active Comparator): 6 cycles before and 6 cycles after surgery consisting in:
  Hour 0: Oxaliplatin 85 mg/m² IV 2-h infusion
  Hour 0: Folinic Acid 400 mg/m² (DL form) or 200 mg/m2 (L form) IV 2-h infusion
  Hour 2: 5-FU 400 mg/m² IV bolus over 2-4 minutes
  Hour 2: 5-FU 2400 mg/m² given as a continuous infusion over 46h.
  On day 1 of a 14 day cycle
  Interventions: Drug: Modified FOLFOX6; Procedure: Surgery
- Arm B: modified FOLFOX6 + Aflibercept and Surgery (Experimental): 6 cycles before and 6 cycles after surgery consisting in:
  Hour 0: Aflibercept 4 mg/kg intravenous infusion 1-h
  Hour 1: Oxaliplatin 85 mg/m2 2-h infusion
  Hour 1: Folinic Acid 400 mg/m2 (DL form) or 200 mg/m2 (L form) 2-h infusion
  Hour 3: 5-FU bolus 400 mg/m2 IV bolus over 2-4 minutes
  Hour 3: 5-FU 2400 mg/m² given as a continuous infusion over 46h.
  Day 1 of a 14 day cycle
  Aflibercept should be given in all cycles, except cycle 6 of pre-operative treatment.
  Interventions: Drug: Modified FOLFOX6; Biological: Aflibercept; Procedure: Surgery

INTERVENTIONS:
Drug: Modified FOLFOX6
  Other Names: 5-FU, folinic acid, oxaliplatin
Biological: Aflibercept — Targeted therapy
  Arms: Arm B: modified FOLFOX6 + Aflibercept and Surgery
Procedure: Surgery

SUMMARY:
Patients presenting with multiple innumerable liver metastases will probably never come to resection, however, for all others, including patients with numerous multiple metastases or large metastases, resection should be considered after limited chemotherapy.

There is consensus for a backbone chemotherapy consisting of fluoropyrimidine + oxaliplatin. FOLFOX was used in the previous EORTC study and is again recommended.

The addition of targeted agents to standard chemotherapy in the perioperative strategy for mCRC might increase the ORR and R0 resectability, without significant increase in toxicity, therefore translating to a better outcome.

BOS2 (EORTC 40091) was designed to test this hypothesis in patients with a KRAS wold-type profile.

It was decided in parallel to design an open label, randomized, multi-center, 2-arm phase II-III study this time aimed at enrolling KRAS mutated patients.

Arm A: (standard) mFOLFOX6 + Surgery Arm B: (experimental) mFOLFOX6 + Aflibercept + Surgery

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CRC with 1 to 8 metachronous or synchronous liver metastases considered to be completely resectable
* Primary tumor (or liver metastasis) of CRC must be KRAS status "mutant"
* Patients must have undergone complete resection (R0) of the primary tumor at least 4 weeks before randomization. Or for patients with synchronous metastases the primary tumor can be resected (R0) at the same time as the liver metastases if: the patient has a non-obstructive primary tumor and is able to receive preoperative chemotherapy (3-4 months) before surgery1.
* Measurable hepatic disease by RECIST version 1.1
* Patients must be 18 years old or older
* A World Health Organization (WHO) performance status of 0 or 1
* Previous adjuvant chemotherapy for primary CRC is allowed if completed at least 12 months before inclusion in this study
* All the following tests should be done within 4 weeks prior to randomization:
* Hematological status: neutrophils (ANC) = 1.5x10 9/L; platelets = 100x10 9/L; haemoglobin = 9g/dL
* Serum creatinine = 1.5 times the upper limit of normal (ULN)
* Proteinuria < 2+ (dipstick urinalysis) or =1g/24hour.
* Liver function: serum bilirubin = 1.5 x upper normal limit (ULN), alkaline phosphatase < 5xULN
* Magnesium ≥ lower limit of normal (LLN)
* Patients with a buffer range from the normal values of +/- 5% for hematology and +/- 10% for biochemistry are acceptable. This will not apply for Renal Function, including Creatinine.
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 14 days prior to the first dose of study treatment.
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Patient should be willing and able to comply with protocol requirements
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Evidence of extra-hepatic metastasis (of CRC)
* Previous chemotherapy for metastatic disease or surgical treatment (e.g. surgical resection or radiofrequency ablation) for liver metastasis. Radiotherapy alone is allowed if given pre or post protocol treatment
* Previous exposure to VEGF/VEGFR targeting therapy within the last 12 months
* Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to randomization
* Gilbert's syndrome
* History of myocardial infarction and/or stroke within 6 months prior to randomization
* Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy
* History or evidence upon physical examination of CNS metastasis
* Bowel obstruction
* Uncontrolled hypercalcemia
* Pre-existing permanent neuropathy (NCI grade = 2)
* Known allergy to any excipient to study drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 1 year
  Increase in progression free survival rate at 1 year in the experimental arm (mFOLFOX6 + aflibercept) compared to mFOLFOX6 alone arm.

SECONDARY OUTCOMES:
Pathological response rate | 4 years
  Increase in major pathological response rate between mFOLFOX6 alone arm and each experimental arm.
Resection rate | 4 years
  Compare the percentage of patients with total resection with these three treatments.
Overall survival | 8 years
  Overall survival is defined as the time interval between the date of randomization and the date of death. Patients who are still alive when last traced will be censored at the date of last follow-up.
Safety | 4 years
  All adverse events will be recorded; the investigator will assess whether those events are drug related (reasonable possibility, no reasonable possibility) and this assessment will be recorded in the database for all adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Nordlinger, Pr., Study Chair — C.H.U. AMBROISE PARE AP-HP, Boulogne-Billancourt, France